CLINICAL TRIAL: NCT02494479
Title: A Randomized, Double Blind, Parallel Group, Placebo Controlled Clinical Study of the Efficacy and Safety of Three Different Daily Dosages of Prurisol Administered Orally to Subjects With Active Mild to Moderate Chronic Plaque Psoriasis
Brief Title: Efficacy and Safety of Prurisol Administered Orally for Active Mild to Moderate Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellceutix Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTIX-PRU-004
Record Dates: First submitted 2015-06-26; First posted 2015-07-10 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2016-05

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Topical Psoriasis; Mild Psoriasis; Moderate Psoriasis; Active Psoriasis; Plaque Psoriasis; Skin Diseases
MeSH Terms: conditions — Psoriasis; Skin Diseases | interventions — abacavir hydroxyacetate; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 50mg of Purisol daily (Active Comparator): One (1) 50 mg tablet of Prurisol and one (1) matching placebo tablet given AM and two (2) matching placebo tablets given PM for 84 (± 3) days
  Interventions: Drug: Prurisol
- 100mg of Purisol daily (Active Comparator): One (1) 50 mg tablets of Prurisol and one (1) matching placebo tablet given twice daily (AM and PM) for 84 (± 3) days
  Interventions: Drug: Prurisol
- 200mg of Purisol daily (Active Comparator): Two (2) 50 mg tablets of Prurisol given twice daily (AM and PM) for 84 (± 3) days
  Interventions: Drug: Prurisol
- Placebo daily (Placebo Comparator): Two (2) placebo tablets given twice daily (AM and PM) for 84 (± 3) days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prurisol — 50mg tablet
  Other Names: Purisol, 50mg tablet
  Arms: 100mg of Purisol daily; 200mg of Purisol daily; 50mg of Purisol daily
Drug: Placebo — Sugar pill designed to match Purisol tablet
  Other Names: Matching Placebo to Purisol tablet
  Arms: Placebo daily

SUMMARY:
This study is designed to evaluate the efficacy and safety of Prurisol using three different oral daily dose regimens administered to subjects with active mild to moderate chronic plaque psoriasis.

DETAILED DESCRIPTION:
The total duration of study participation for an individual subject is approximately 112 days (16 weeks) consisting of a Screening visit, followed within 21 days by Randomization and a Treatment Period of 84 days, and a Follow-up Period of 28 days after the last day of study drug treatment. A window of ± 3 days will be considered acceptable for conduct of each scheduled visit following the first visit.

This study will require eight (8) scheduled subject visits:

x Visit 1: Screening (Up to Day 21) x Visit 2: Baseline (Day 0) x Visit 3: Day 14 Interim (± 3 days) x Visit 4: Day 28 Interim (± 3 days) x Visit 5: Day 42 Interim (± 3 days) x Visit 6: Day 56 Interim (± 3 days) x Visit 7: Day 84 End of Treatment/Unscheduled/ET (± 3 days) x Visit 8: Day 112 Follow-up (± 3 days)

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female adults aged 18 years with a clinical diagnosis of stable (at least 6 months) plaque psoriasis, not including scalp or intertriginous areas.
* The extent of psoriasis must meet all of the following three (3) criteria:

  * Total Body Surface Area (BSA) affected by plaque psoriasis of 10% to 20% inclusive
  * Investigator's Global Assessment (IGA) score of the severity of psoriasis of 2 or 3 (5- point ordinal scale)
  * Identification of a target psoriatic lesion with a score of 3 on the Target Lesion Assessment scale (5-point ordinal scale) for Scaling. (Other psoriatic lesions may have lower scaling scores.)
* Females of reproductive potential must not be pregnant
* Female subjects with reproductive potential, if sexually active, must agree to use reliable means of contraception
* The subject must agree to avoid prolonged exposure to the sun and avoid the use of tanning booths or other ultraviolet light sources during the study.
* The subject must provide signed and dated written informed consent to participate in the clinical study.

Exclusion Criteria:

* 1. Females of reproductive potential who are not using reliable contraception.
* Presence of any non-psoriatic uncontrolled (in the Investigator's medical opinion) systemic disease. i
* Unstable forms of psoriasis, e.g. guttate, erythrodermic, exfoliative, palmoplantar, nail, or pustular.
* Use within 6 months of biologic treatment for psoriasis
* Use within 24 months of chemotherapy or radiation therapy.
* Use within 2 months of any systemic immunosuppressive therapy.
* Use within 1 month of (1) systemic corticosteroids, (2) systemic antibiotics, (3) systemic antipsoriasis treatments (e.g. methotrexate, corticosporin, hydroxyurea), (4) PUVA therapy, (5) UVB, (6) systemic anti-inflammatory treatment.
* Use within 2 weeks of topical antipsoriasis drugs or topical corticosteroids or topical retinoids.
* Presence of a condition (e.g., history of frequent consumption of substantial quantities of alcohol, or an untreated psychiatric condition) that makes it unlikely that the requirements of the protocol will be completed.
* History of any previous use of a Tumor Necrosis Factor (TNF) blocker or other immunomodulating drug as therapy for psoriasis within the 6 months prior to screening.
* History of any allergic reaction to any formulation of abacavir.
* Previous treatment with any abacavir-containing product, e.g., Ziagen®, Epzicom®, or Trizivir®.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the percentage of subjects with ≥ 2 point improvement in IGA rating as defined by visual inspections of patient lesions | 84 days

SECONDARY OUTCOMES:
The Secondary efficacy endpoints are the percentage of subjects in each treatment group with:≥ 2 point improvement in IGA at 28 days | 28 days
The Secondary efficacy endpoints are the percentage of subjects in each treatment group with: ≥ 2 point improvement in IGA at 56 days | 56 Days
The Secondary efficacy endpoints are the percentage of subjects in each treatment group with: ≥1 point improvement in Scaling Score of Target Lesion at 28 days | 28 Days
The Secondary efficacy endpoints are the percentage of subjects in each treatment group with: ≥1 point improvement in Scaling Score of Target Lesion at 56 days | 56 Days
The Secondary efficacy endpoints are the percentage of subjects in each treatment group with: ≥1 point improvement in Scaling Score of Target Lesion at 84 days | 84 Days

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Cellceutix Study Center, Huntsville, Alabama
  - Cellceutix Study Center, Encino, California
  - Cellceutix Study Center, Coral Gables, Florida
  - Cellceutix Study Center, Hialeah, Florida
  - Cellceutix Study Center, Kissimmee, Florida
  - Cellceutix Study Center, Miami, Florida
  - Cellceutix Study Center, Pembroke Pines, Florida
  - Cellceutix Study Center, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No